CLINICAL TRIAL: NCT06135285
Title: Korus: Smart Mattress to Prevent Night-time Sudden Unexpected Death in Epilepsy (SUDEP)
Brief Title: Korus: a Device to Prevent Sudden Unexpected Death in Epilepsy (SUDEP)
Acronym: Korus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jong Woo Lee, Associate Professor of Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2023P002023
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Control subjects (Experimental): The subject will lie down on the Korus smart mattress. Korus will detect when the subject is in a prone (face-down) position and reposition the subject into a recovery (sideways) position.
  Interventions: Device: Control subjects

INTERVENTIONS:
Device: Control subjects — The subject will be repositioned from the prone to recovery position

SUMMARY:
The goal of this feasibility study is to test the Korus smart mattress in healthy volunteers. The main questions it aims to answer are:

* Can Korus accurately detect body position in bed (left, right, supine, prone)
* Can Korus reposition the subject from a prone to recovery (sideways) position? Participants will be asked to lie down on Korus and turn into various positions; when the prone position is detected, they will be repositioned.

DETAILED DESCRIPTION:
Korus is a a smart mattress consisting entirely of pneumatically inflatable smartcells with embedded sensors. It is designed to detect a subject's body position an inflate the proper smartcells to reposition a subject from the prone to the recovery (sideways) position. Healthy control subjects will be recruited to test Korus' sensing system and its performance in repositioning the subject. Korus will utilize specialized sensors and a computer learning algorithm to detect the subject's body position. Based on this data, Korus will activate the appropriate smart cells to reposition the subject.

ELIGIBILITY:
Inclusion Criteria:

• Adults age 18-65; at least 30% of subjects will be self-identified as prone sleepers

Exclusion Criteria: any significant medical history for which body movements will potentially be harmful, including but not limited to:

* History of neurological dysfunction, including spinal cord abnormalities
* History of psychiatric disorder, including anxiety
* History of cardiac dysfunction
* History of osteoporosis or osteopenia
* History of significant orthopedic dysfunction
* History of falls
* History of sleep disorder
* Taking neuroactive medications
* Taking anticoagulants
* Current recreational drug use
* BMI under 18 or over 30
* Systolic BP >180 or <90
* Open wounds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Body position detection | 5 seconds
  Correct detection of one of 4 cardinal body positions: prone, supine, left, right
Number of subjects correctly repositioned from the prone to recovery position | 30 seconds
  We will measure the performance of Korus to successfully reposition the subject from the prone to recovery position

CONTACTS AND LOCATIONS:
Overall Officials: Jong Woo Lee, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will collect and generate the following data from 50 normative control subjects: a) spontaneous body position as recorded by the KORUS sensor; b) subject demographics: age, sex, height, weight
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be deposited starting 12 months after the study completion
Access Criteria: To request access of the data, researchers will use the standard processes at PhysioNet, where the data will be stored, which will decide which requests to grant.

REFERENCES:
- [Background] Ryvlin P, Nashef L, Lhatoo SD, Bateman LM, Bird J, Bleasel A, Boon P, Crespel A, Dworetzky BA, Hogenhaven H, Lerche H, Maillard L, Malter MP, Marchal C, Murthy JM, Nitsche M, Pataraia E, Rabben T, Rheims S, Sadzot B, Schulze-Bonhage A, Seyal M, So EL, Spitz M, Szucs A, Tan M, Tao JX, Tomson T. Incidence and mechanisms of cardiorespiratory arrests in epilepsy monitoring units (MORTEMUS): a retrospective study. Lancet Neurol. 2013 Oct;12(10):966-77. doi: 10.1016/S1474-4422(13)70214-X. Epub 2013 Sep 4. PMID 24012372
- [Background] Tao JX, Sandra R, Wu S, Ebersole JS. Should the "Back to Sleep" campaign be advocated for SUDEP prevention? Epilepsy Behav. 2015 Apr;45:79-80. doi: 10.1016/j.yebeh.2015.02.020. Epub 2015 Apr 11. No abstract available. PMID 25875185